CLINICAL TRIAL: NCT00248300
Title: A Peri-intubation Oral Intervention to Reduce Oral Flora and VAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Uniformed Services University of the Health Sciences (U.S. Federal Agency); TriService Nursing Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SToPP-IT; MDA-905-03-1-TS02, N03-006
Record Dates: First submitted 2005-11-01; First posted 2005-11-03 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Pneumonia
Keywords: ventilator-associated pneumonia; hospital acquired pneumonia
MeSH Terms: conditions — Pneumonia; Pneumonia, Ventilator-Associated; Healthcare-Associated Pneumonia | interventions — Chlorhexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Chlorhexidine — Chlorhexidine, 5 ml swab to the oral cavity within 12 hours of endotracheal tube intubation

SUMMARY:
The purpose of this study is determine if a single, early dose of chlorhexidine applied within 12 hours after endotracheal tube insertion will reduce the bacteria in the oral cavity and the incidence of pneumonia in trauma victims.

DETAILED DESCRIPTION:
Pneumonia is the leading cause of death from nosocomial infections. Intubation and mechanical ventilation greatly increase the risk of ventilator associated pneumonia (VAP) which is highest in trauma, burn, neurosurgical and surgical patients. Oral bacteria have been shown to be responsible for the development of VAP since the endotracheal tube provides a pathway for direct entry of bacteria from the oropharynx to the respiratory tract. Therefore, reducing the number of microorganisms in the mouth reduces the pool of organisms available for translocation to and colonization of the lung. The Tri-Service Oral Health Survey showed that military recruits had inferior oral health when compared to their civilian cohorts. Further, oral hygiene is likely to deteriorate in combat situations, increasing oral microbial flora. Intubation of combat casualties in the future will likely be performed in the field by the EMT-B trained combat medic (91W) under adverse conditions. Therefore, interventions to reduce oral microbial flora with intubation are attractive to reduce the incidence of VAP in combat casualties. This study will test the effect of a single peri-intubation oral intervention on oral microbial flora and the development of VAP in traumatic injury. Two hundred trauma patients requiring endotracheal intubation will be randomly assigned to either the intervention or control group over an 18-month data collection period. Data related to oral microbial flora (measured by semi-quantitative oral culture) and VAP (measured by the clinical pulmonary infection score-CPIS) will be obtained on study admission, at 24 (oral culture data only), 48 and 72 hours after intubation. The exact Wilcoxon two-sample one-sided test will be used to test for difference between groups. CPIS data will be compared using an analysis of covariance model. Covariates such as baseline oral culture category, trauma-injury and severity score (TRISS), illness severity (APACHE III) and frequency and timing of usual oral care will also be included. The findings from this study will be the first report of an empirically based peri-intubation oral intervention to reduce VAP and can be easily applied to the care of traumatic injury in both combat and civilian casualties.

ELIGIBILITY:
Inclusion Criteria:

* trauma victim
* endotracheal intubation within the past 12 hours
* mechanical ventilation

Exclusion Criteria:

* diagnosis of pneumonia at the time of intubation
* previous endotracheal tube placement in the last 48 hours
* burn injuries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2005-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Oral microbial flora -- measured by semi-quantitative oral culture | At 24, 48 and 72 hours after intubation

SECONDARY OUTCOMES:
Incidence of ventilator associated pneumonia, measured by the clinical pulmonary infection score (CPIS) and obtained on study admission, 48 and 72 hours after intubation | At 48 and 72 hours after intubation.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jo E Grap, PhD, Principal Investigator — Virginia Commonwealth University School of Nursing
Locations (1):
- Virginia Commonwealth University School of Nursing, Richmond, Virginia, United States

REFERENCES:
- [Background] Grap MJ, Munro CL, Elswick RK Jr, Sessler CN, Ward KR. Duration of action of a single, early oral application of chlorhexidine on oral microbial flora in mechanically ventilated patients: a pilot study. Heart Lung. 2004 Mar-Apr;33(2):83-91. doi: 10.1016/j.hrtlng.2003.12.004. PMID 15024373